CLINICAL TRIAL: NCT03522974
Title: Effects of Freeze Dried Strawberry Powder Supplementation on Vascular Function, Blood Markers of Cardiovascular Risk, and the Gut Microbiome
Brief Title: Effects of Freeze Dried Strawberry Powder Supplementation on Cardiovascular Risk Factors and Gut Microbiome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID stopped clinical research trials and industry pulled funding
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Ann Skulas-Ray, Assistant Professor of Nutritional Sciences, University of Arizona
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Strawberry Study
Record Dates: First submitted 2018-04-30; First posted 2018-05-14 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Cardiovascular Risk Factor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): 40 g/d placebo powder
  Interventions: Dietary Supplement: Placebo powder
- Strawberry powder (high dose) (Experimental): 40 g/d freeze dried strawberry powder
  Interventions: Dietary Supplement: Strawberry powder
- Strawberry powder (low dose) (Active Comparator): 13 g/d freeze dried strawberry powder
  Interventions: Dietary Supplement: Strawberry powder

INTERVENTIONS:
Dietary Supplement: Strawberry powder — Freeze dried strawberry powder
  Arms: Strawberry powder (high dose); Strawberry powder (low dose)
Dietary Supplement: Placebo powder — 40 g/d placebo powder matched for taste and appearance
  Arms: Placebo

SUMMARY:
Dietary interventions designed to promote health by increasing the consumption of particular health-promoting foods (e.g., strawberries) generally target blood pressure and LDL-C; however, CVD risk reduction may also be achieved via changes in emerging endpoints such as the gut microbiome. Previous research suggests that strawberries have the potential to reduce LDL-C, but it remains unclear whether there is a dose-response relationship. Moreover, few studies have evaluated effects on vascular health or characterized changes in the gut microbiome following daily strawberry consumption. Additionally, previous studies have largely been conducted among Caucasian populations. Given the demographics of the US, it is important to evaluate effects in study populations that include ethnicities that may have higher risk of type 2 diabetes and/or other CVD risk factors, such as Hispanics. This study aims to examine the effects of 4 weeks of supplementation with two doses of freeze dried strawberry powder (low dose: 13 g/d and high dose: 40 g/d) on: 1) LDL-C and blood pressure; 2) gut microbiome profile; and 3) other CVD and type 2 diabetes risk factors, including glucose, insulin, and inflammatory markers. Overweight (BMI 25-36 kg/m2) but otherwise healthy adults with moderately elevated LDL-C (>3.0 mmol/L) and/or prehypertension (120-159/80-99 mm Hg) will be enrolled. This will optimize the potential for observing significant benefits on these outcomes. 50 eligible participants will be recruited with the expectation that at least 40 will complete the study. The placebo-controlled, crossover study design will allow for a direct comparison of dose-response within the same participant. The investigators anticipate that the bioactive components of strawberries will reduce LDL-C and blood pressure, and modify the gut microbiome, with greater changes on the high dose. There is preliminary evidence that polyphenol-rich foods can modify gut microbiota profiles, but this would be the first study to characterize the effects of daily strawberry consumption. The investigators are uniquely placed at the University of Arizona to enroll a larger percentage of Hispanic participants, who are often under-represented in clinical nutritional research. Results from the proposed study will improve understanding of how strawberries might promote health, and could provide further support for the incorporation of whole freeze dried fruit in dietary guidelines.

ELIGIBILITY:
Inclusion Criteria:

* At least one of the following:

  * LDL-C above 3.0 mmol/L (116 mg/dL)
  * Systolic blood pressure of 120-159 mmHg
  * Diastolic blood pressure of 80-99 mmHg
* Total cholesterol below 6.2 mmol/L (240 mg/dL)
* Triglycerides below 350 mg/dL

Exclusion Criteria:

* Allergies to strawberries
* History of CVD, Stage II hypertension (BP ≥ 160/100 mmHg), kidney disease, diabetes, or inflammatory diseases such as GI disorders and rheumatoid arthritis
* Use of medications/supplements for elevated lipids, blood pressure, or glucose
* Chronic use of non-steroidal anti-inflammatory or immunosuppressant drugs
* Conditions requiring chronic use of steroids

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
LDL-C/non-HDL-C | 4-6 weeks
Brachial and central blood pressure | 4-6- weeks
  systolic and diastolic blood pressures

SECONDARY OUTCOMES:
Pulse Wave Velocity (PWV) | 4-6 weeks
Augmentation Index | 4-6 weeks
  augmentation index corrected for heart rate
Other lipids and lipoproteins | 4-6 weeks
  HDL-C, total cholesterol, and triglycerides
Glucose | 4-6 weeks
  fasting glucose
Insulin | 4-6 weeks
  fasting insulin

OTHER OUTCOMES:
Gut microbiome | 4-6 weeks
  Composition of the gut microbial community measured by high-throughput 16S rRNA sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] U.S. Department of Health and Human Services and U.S. Department of Agriculture, 2015-2020 Dietary Guidelines for Americans, 2015.
- [Background] Basu A, Betts NM, Nguyen A, Newman ED, Fu D, Lyons TJ. Freeze-dried strawberries lower serum cholesterol and lipid peroxidation in adults with abdominal adiposity and elevated serum lipids. J Nutr. 2014 Jun;144(6):830-7. doi: 10.3945/jn.113.188169. Epub 2014 Mar 26. PMID 24670970
- [Background] Jennings A, Welch AA, Fairweather-Tait SJ, Kay C, Minihane AM, Chowienczyk P, Jiang B, Cecelja M, Spector T, Macgregor A, Cassidy A. Higher anthocyanin intake is associated with lower arterial stiffness and central blood pressure in women. Am J Clin Nutr. 2012 Oct;96(4):781-8. doi: 10.3945/ajcn.112.042036. Epub 2012 Aug 22. PMID 22914551
- [Background] Tuohy KM, Conterno L, Gasperotti M, Viola R. Up-regulating the human intestinal microbiome using whole plant foods, polyphenols, and/or fiber. J Agric Food Chem. 2012 Sep 12;60(36):8776-82. doi: 10.1021/jf2053959. Epub 2012 Jun 12. PMID 22607578
- [Background] Richter CK, Skulas-Ray AC, Gaugler TL, Lambert JD, Proctor DN, Kris-Etherton PM. Incorporating freeze-dried strawberry powder into a high-fat meal does not alter postprandial vascular function or blood markers of cardiovascular disease risk: a randomized controlled trial. Am J Clin Nutr. 2017 Feb;105(2):313-322. doi: 10.3945/ajcn.116.141804. Epub 2016 Dec 21. PMID 28003205
- [Background] Burton-Freeman B, Linares A, Hyson D, Kappagoda T. Strawberry modulates LDL oxidation and postprandial lipemia in response to high-fat meal in overweight hyperlipidemic men and women. J Am Coll Nutr. 2010 Feb;29(1):46-54. doi: 10.1080/07315724.2010.10719816. PMID 20595645
- [Background] Zunino SJ, Parelman MA, Freytag TL, Stephensen CB, Kelley DS, Mackey BE, Woodhouse LR, Bonnel EL. Effects of dietary strawberry powder on blood lipids and inflammatory markers in obese human subjects. Br J Nutr. 2012 Sep;108(5):900-9. doi: 10.1017/S0007114511006027. Epub 2011 Nov 9. PMID 22068016
- [Background] Park E, Edirisinghe I, Wei H, Vijayakumar LP, Banaszewski K, Cappozzo JC, Burton-Freeman B. A dose-response evaluation of freeze-dried strawberries independent of fiber content on metabolic indices in abdominally obese individuals with insulin resistance in a randomized, single-blinded, diet-controlled crossover trial. Mol Nutr Food Res. 2016 May;60(5):1099-109. doi: 10.1002/mnfr.201500845. Epub 2016 Mar 29. PMID 26842771
- [Background] Erlund I, Koli R, Alfthan G, Marniemi J, Puukka P, Mustonen P, Mattila P, Jula A. Favorable effects of berry consumption on platelet function, blood pressure, and HDL cholesterol. Am J Clin Nutr. 2008 Feb;87(2):323-31. doi: 10.1093/ajcn/87.2.323. PMID 18258621
- [Background] Vendrame S, Guglielmetti S, Riso P, Arioli S, Klimis-Zacas D, Porrini M. Six-week consumption of a wild blueberry powder drink increases bifidobacteria in the human gut. J Agric Food Chem. 2011 Dec 28;59(24):12815-20. doi: 10.1021/jf2028686. Epub 2011 Nov 18. PMID 22060186
- [Background] Espin JC, Larrosa M, Garcia-Conesa MT, Tomas-Barberan F. Biological significance of urolithins, the gut microbial ellagic Acid-derived metabolites: the evidence so far. Evid Based Complement Alternat Med. 2013;2013:270418. doi: 10.1155/2013/270418. Epub 2013 May 28. PMID 23781257

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT03522974/Prot_SAP_001.pdf
  • Informed Consent Form (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT03522974/ICF_000.pdf